CLINICAL TRIAL: NCT04464668
Title: Colorectal Cancer Awareness, Research and Education and Screening - Rural Expansion, Access and Capacity for Health
Acronym: CARES-REACH
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-20560
Record Dates: First submitted 2020-07-02; First posted 2020-07-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: Fecal Immunochemical Test; F.I.T.
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Wave 1 Only: Clinics using CARES Intervention: Based on a stratified (rural vs urban) procedure, investigators will randomly select 7 clinics to implement the Colorectal Cancer Awareness, Research, Education & Screening (CARES) intervention.
  Interventions: Behavioral: Provider Tools; Behavioral: Provider surveys
- Wave 1 Only: Control Clinics: Based on a stratified (rural vs urban) procedure, investigators will randomly select 7 clinics as control (usual care) clinics.
- All Clinics: For Wave 2, the 7 clinics in the control group will roll out as intervention clinic, thus, all 14 clinics will be exposed to the intervention by year 2.
  Interventions: Behavioral: Provider Tools; Behavioral: Provider surveys

INTERVENTIONS:
Behavioral: Provider Tools — Providers will be trained to use Electronic Medical Record (EMR) tools and prompts, and an organization wide cancer control champion will be trained to motivate providers and navigate patients.
  Groups: All Clinics; Wave 1 Only: Clinics using CARES Intervention
Behavioral: Provider surveys — Remote/electronic data collection surveys will be conducted with clinic institution leaders, cancer control champions, and providers from various clinic locations to solicit feedback about implementation processes at three time points (baseline, mid-point and end of study implementation)
  Groups: All Clinics; Wave 1 Only: Clinics using CARES Intervention

SUMMARY:
This study is to assess the impact of the CARES-REACH intervention on colorectal cancer screening rates.

DETAILED DESCRIPTION:
This study will not accrue individual patients. Instead, the investigators are collecting process data from health care providers to determine the procedures that impact or help to increase colorectal cancer screening rates.

ELIGIBILITY:
Inclusion Criteria:

* Staff and providers working in a clinic within one of the two participating systems
* Involved in adult patient care

Exclusion Criteria:

* Staff and providers who are not engaged in directing or decisions related to colo-rectal cancer screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff and providers from the two participating Federally Qualified Health Care systems - Central Florida Health Centers and Manatee County Rural Health Services.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2027-10-26 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Colorectal Cancer Screening Rates - Initial FIT | Years 1-5
  Percentage of patients who complete initial Fecal Immunochemical Test (FIT)
Change in Colorectal Cancer Screening Rates - Repeat FIT | Years 1-5
  Percentage of patients who complete a repeat Fecal Immunochemical Test (FIT)

SECONDARY OUTCOMES:
Differences in Screening Rates | Years 2-5
  Screening rate differences to determine how variables such as clinic setting (rural vs urban), population characteristics such as nativity (foreign born status), language preference, education, income, health insurance, etc. differentially impact annual clinic Colorectal Cancer (CRC) screening rates.

CONTACTS AND LOCATIONS:
Overall Officials: Clement K Gwede, PhD MPH RN FAAN, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- [Derived] Montoya SM, Olaore P, Bastardo-Acosta J, Abdulla R, Schell MJ, Hidalgo A, Turner B, Rider M, Kishun-Jit N, Joshua A, Pollard J, Friedman M, Christy SM, Meade CD, Gwede CK. Protocol paper for an implementation science approach to promoting colorectal cancer screening in Federally Qualified Health Center clinics: A stepped-wedge, multilevel intervention trial. Res Sq [Preprint]. 2024 Jul 18:rs.3.rs-4558718. doi: 10.21203/rs.3.rs-4558718/v1. PMID 39070625